CLINICAL TRIAL: NCT05974722
Title: A Randomized, Blinded, Parallel-group Trial Evaluating Mesh Versus Pledgeted Sutures in Paraesophageal Hernia Recurrence
Brief Title: Mesh Vs Pledgets for Repair of Paraesophageal Hernia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: David Krpata (Other)
Responsible Party: Sponsor-Investigator, David Krpata, Professor of Surgery, CCF Lerner College of Medicine, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 22-1109
Record Dates: First submitted 2023-07-15; First posted 2023-08-03 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-07

CONDITIONS: Paraesophageal Hernia; GERD
MeSH Terms: conditions — Hernia, Hiatal; Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive mesh or pledgeted suture reinforcement of the crural repair
Who Masked: Participant, Care Provider
Masking Description: Patients will be blinded to the intervention. Additionally, there will be blinded outcome assessors/study team including 3 surgeons reviewing recurrence imaging
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Mesh-based crural reinforcement (Other): Patient will receive Ovitex mesh to reinforce the crural repair
  Interventions: Device: OviTex Mesh
- Pledgeted suture-based crural reinforcement (Other): Patient will receive pledgeted sutures to reinforce the crural repair
  Interventions: Other: Pledgeted sutures

INTERVENTIONS:
Device: OviTex Mesh — Patient will receive Ovitex Mesh (TELA Bio)
  Arms: Mesh-based crural reinforcement
Other: Pledgeted sutures — Patient will receive pledgeted sutures
  Arms: Pledgeted suture-based crural reinforcement

SUMMARY:
The goal of this clinical trial is to compare whether the use of Ovitex mesh provides superior reduction in 2-year recurrence compared to pledgeted suture closure (no mesh) for patients undergoing paraesophageal hernia repair at the Cleveland Clinic. The main questions it aims to answer are:

* Determine whether there is a difference in 2-year rates of radiographic recurrence with Ovitex versus pledgeted sutures in paraesophageal hernia repair.
* Assess patient quality of life (QOL) after paraesophageal hernia repair with pledgets and mesh. A two-tailed research hypothesis will be used to determine whether there are differences between the two arms

DETAILED DESCRIPTION:
This is a prospective, single-center, randomized, two-arm trial assessing the impact of Ovitex mesh on paraesophageal hernia recurrence. This study will occur at Cleveland Clinic Foundation in Cleveland, OH. A total of 164 patients will be enrolled in this study. The anticipated accrual rate is approximately 7 per month for a total accrual period of approximately 24 months.

Patients may be enrolled into the study provided all inclusion and no exclusion criteria are met as specified in Section 4. Subjects will be evaluated through hospital discharge and return for follow-up visits at 1 month (10 days-45 days) and annually through 2 years postoperatively. Total estimated duration for the trial is 4 years for the primary outcome with an additional 3 years for longer term follow up resulting in a total of 7 years.

Several approaches to limiting bias are included in this trial.

* Intraoperative bias- limited by randomization just prior to crural closure
* Blinded outcome assessors/study team including 3 surgeons reviewing recurrence imaging
* Single blind - patients blinded to intervention Devices included in this study include Ovitex mesh and pledgets which are both used to reinforce the repair at the crura. Ovitex mesh is FDA approved for this indication.

Study Endpoints Primary Endpoint The primary endpoint of this study is the binary 2-year rate of radiographic recurrence of the paraesophageal hernia, defined gastroesophageal junction at least 2 cm above the hiatus on upper GI studies, CT, or MRI. Anatomical recurrence assessed via imaging is the gold standard of diagnosing recurrence, and thus is the most appropriate primary outcome.

Secondary Endpoints

* Patient quality of life (measured at baseline, 30 days, and annually)

  * EQ5D
  * EQ-VAS
  * Decision regret index (only measured annually)
  * GERD-HRQL
  * Presence of regurgitation, chest pain, abdominal pain, nausea, vomiting, postprandial pain, cardiovascular, and pulmonary symptoms
* Immediate recurrence rates (within 45 days of surgery)
* Reoperation rates throughout the study
* Cost
* Safety endpoints:

  * Intraoperative complications: solid organ injury, etc.
  * Clavien-Dindo complications
  * Comprehensive Complications Index
  * Foregut complications requiring re-interventions

While anatomic recurrence is extremely important from a surgical perspective, patients often have variable impacts of recurrence on quality of life. Furthermore, there is significant variability in symptoms for patients with recurrence. These secondary outcomes will help us to characterize the impact of potential recurrences on the patient.

Additionally, immediate recurrences offer insight into possible issues with the repair and are important to evaluate. Rates of reoperation can indicate the severity of the recurrence's impact on quality of life. Given the concerns about mesh complications, safety endpoints are necessary. Since the use of mesh is more expensive than not using mesh, collecting data on cost will help in future cost effectiveness analyses.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Willing and able to provide informed consent
* Willing and able to participate in long-term follow up including study visits and surveys
* Type II, III, or IV hiatal hernia > 5 cm, confirmed via upper GI studies, CT, or MRI 5 cm or greater hernia confirmed intraoperatively

Exclusion Criteria:

* Pregnancy
* BMI >45
* Allergy to any components of mesh
* Patients undergoing PEHR with a concurrent bariatric procedure or other procedure to reduce stomach volume (sleeve gastrectomy, roux-en-y gastric bypass, duodenal switch, single-anastomosis gastric bypass, and partial or total gastrectomy)
* Patients who have undergone previous hiatal hernia repair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Radiographic recurrence rate | 2 years after surgery
  The primary endpoint of this study is the binary 2-year rate of radiographic recurrence of the paraesophageal hernia, defined gastroesophageal junction at least 2 cm above the hiatus on upper gastrointestinal studies, CT, or MRI.

SECONDARY OUTCOMES:
Patient quality of life as measured by the validated EQ5D survey | Preop, 30-day, 1-year, and 2-year timepoints after surgery
  Patient quality of life will be assessed using the validated EQ5D (EuroQol 5 Dimension) survey measuring self-reported assessments of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression between the two groups.
Patient quality of life as measured by the validated EQ-VAS survey | Preop, 30-day, 1-year, and 2-year timepoints after surgery
  Patient quality of life will be assessed using the validated EQ-VAS (EuroQol Visual Analog Scale) that takes values between 100 (best imaginable health) and 0 (worst imaginable health), on which patients provide a global assessment of their health attributed by paraesophageal hernias and compared between the two groups. This scale was designed to be used in conjunction with the EQ5D survey.
Patient quality of life as measured by the validated decision regret scale survey | 1-year, and 2-year timepoints after surgery
  Patient quality of life will be assessed using the validated decision regret scale, a 5-item survey used to serve as an indicator of health care decision regret at a given point in time attributed by undergoing surgery for the patient's paraesophageal hernia and compared between the two groups. The patients are asked 5 questions regarding the decision to undergo the surgery and to indicate the extent to which they agree or disagree with the statements in the regret scale by indicating a number from 1 (Strongly Agree) to 5 (Strongly Disagree) that best indicates their level of agreement. To obtain a final score, the items are converted to a 0-100 scale by subtracting 1 from each item then multiplying by 25. A score of 0 means no regret; a score of 100 means high regret. Final scores will be compared between the two groups.
Patient quality of life as measured by the GERD-HRQL scale | Preop, 30-day, 1-year, and 2-year timepoints after surgery
  Patient quality of life will be assessed using the validated GERD-HRQL (GastroEsophageal Reflux Disease Health-Related Quality of Life) scale, which provides a quantitative method of measuring GERD symptoms severity and contains a total of 10 scaled items (Likert 0-5, with higher score indicating worse symptoms). A minimum composite score of 0 will be the best possible score (asymptomatic in all items) and the maximum score of 50 represents incapacitation in all items. Composite scores will be compared between the two groups.
Patient satisfaction as measured by patient reported assessment | Preop, 30-day, 1-year, and 2-year timepoints after surgery
  Patient-reported global satisfaction assessment within the GERD-HRQL (GastroEsophageal Reflux Disease Health-Related Quality of Life) survey. The patient will answer whether they are satisfied, neutral, or dissatisfied with their present condition at the time of completing the GERD-HRQL. Their answers will be interpreted as a patient-reported 'global' assessment of their condition with respect to GERD and compared between the two groups.
Patient quality of life as measured by presence of patient reported dysphagia symptoms | Preop, 30-day, 1-year, and 2-year timepoints after surgery
  A dysphagia scale will be used to measure the presence of 8 symptoms (regurgitation, chest pain, abdominal pain, nausea, vomiting, postprandial pain, cardiovascular, and pulmonary symptoms) over the prior 7 days, each on a 0-10 scale with 0 representing "no effect on life" and 10 representing "extreme effect on life." Mean scores for each symptom will be compared between the two groups.
Immediate recurrence | Within 45 days from surgery
  The rates of immediate paraesophageal recurrence (as defined as within 45 days of surgery) will be compared between the 2 groups.
Reoperations | Throughout study up to 2 years after surgery
  Reoperation rates for paraesophageal hernia will be compared between the two groups throughout the study
Intraoperative complications | At time of surgery
  Intraoperative complications (solid organ injury, etc.) will be recorded and compared between the two groups.
Clavien-Dindo Complications | Throughout study up to 2 years after surgery
  The Clavien-Dindo complication classification, which consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb, and V) where higher grades mean increased severity of complication, will be used to categorize complications for each patient and compared between the two groups.
Comprehensive Complications Index (CCI) | Throughout study up to 2 years after surgery
  The Comprehensive Complications Index (CCI), which is calculated as the sum of all complications and weighted for their severity based on the Clavien-Dindo classification will be calculated for each patient and compared between the two groups. The CCI scale ranges from 0 (no complication) to 100 (death).
Foregut complications requiring reintervention | Throughout study up to 2 years after surgery
  Foregut complications requiring reinterventions will be recorded for each patient and compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: David M Krpata, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Center for Abdominal Core Health, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No